CLINICAL TRIAL: NCT05675020
Title: Promote Healthy Lifestyle Behaviors for Adolescents With Mental Health Conditions
Brief Title: Promoting Healthy Lifestyle Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Rachel Sharp, Principal Investigator, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003072
Record Dates: First submitted 2022-12-14; First posted 2023-01-09 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Behavioral / Psychiatric Disorder; Lifestyle, Healthy
Keywords: Adolescent; Behavioral Health Condition; Behavioral / Psychiatric Disorder; Lifestyle Modification; Lifestyle; Healthy
MeSH Terms: conditions — Behavior; Mental Disorders

STUDY DESIGN:
Intervention Model Description: * This project utilizes a one-group pretest-posttest design study for 9 adolescents (aged 12-17 years) diagnosed with a mental health condition(s) and their parent/legal guardian.
  * This educational program will be delivered via a 45-minute presentation via Zoom.
  * Participants will have the option to select between multiple dates and times for educational presentation
  * The educational presentation will be recorded and emailed to participants within 1 week of intervention to re-watch/review.
  * The educational program will promote healthy lifestyle knowledge and behaviors through education evidenced by the Centers for Disease Control (CDC), World Health Organization (WHO), and the American Academy of Pediatrics.
  * We will compare the effects of an educational program on healthy lifestyle knowledge and behaviors pre-and post-program (after one month) via a REDCap survey for the adolescent and their parent/legal guardian.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent-Adolescent Dyad (Experimental): Each parent-adolescent dyad will receive the intervention (educational program delivered via a 45-minute presentation via Zoom).
  The educational program will promote healthy lifestyle knowledge and behaviors through education evidenced by the CDC, WHO, and the American Academy of Pediatrics. Educational sessions will include the importance of healthy lifestyle modifications in the adolescent population with a mental health condition(s), lifestyle recommendations versus reality, nutrition, physical activity, screen time, and sleep recommendations and guidelines. The educational presentation will include 5-10 minutes of education regarding recommendations versus reality for nutrition, PA, screen time, and sleep, 20-25 minutes of education regarding ways to improve healthy lifestyle knowledge and behaviors, 10 minutes for questions and discussion.
  Interventions: Behavioral: Zoom Intervention

INTERVENTIONS:
Behavioral: Zoom Intervention — This educational program will be delivered via a 45-minute presentation via Zoom.
  * The educational presentation will be recorded and emailed to participants within 1 week of intervention to re-watch/review.
  * The educational program will promote a healthy lifestyle knowledge and behaviors through education evidenced by the CDC, WHO, and the American Academy of Pediatrics. Educational sessions will include the importance of healthy lifestyle modifications in the adolescent population with a mental health condition(s), lifestyle recommendations versus reality, nutrition, physical activity, screen time, and sleep recommendations and guidelines.
  * We will compare the effects of an educational program on healthy lifestyle knowledge and behaviors pre-and post-program (after one month) via a REDCap survey for the adolescent and their parent/legal guardian.

SUMMARY:
This study's purpose is to identify factors that may aid in answering the clinical question: Among adolescents 12-17 years old who are diagnosed with a mental health condition(s), does a family-based educational intervention improve healthy lifestyle knowledge and behaviors, including nutrition, PA, screen time, and sleep? The specific aims are to: Aim 1: To educate adolescents with mental health conditions and their family members about ways to improve healthy lifestyle behaviors. Aim 2: To evaluate an increase in knowledge on healthy lifestyle behaviors after a 45-minute online education session. Aim 3: To evaluate an increase in healthy lifestyle behaviors after the intervention.

This project utilizes a one-group pretest-posttest design study for 30 adolescents (aged 12-17 years) diagnosed with a mental health condition(s) and their parent/legal guardian. This project will implement best practices to promote healthy lifestyle knowledge and behaviors to adolescents and their parent(s)/legal guardian(s). This will be a 45-minute educational presentation delivered via Zoom. Participants will have option to select between 2-3 dates and times for educational presentation. The investigators will compare the effects of an educational program on healthy lifestyle knowledge and behaviors pre-and post-program (after one month) via a REDCap survey for the adolescent and their parent/legal guardian. The survey will utilize an adapted version of the 2021 National Youth Risk Behavior Survey (YRBS) and the 2020 National Survey of Children's Health (NSCH-T3). The analysis of this project will compare changes in healthy lifestyle knowledge and behaviors using a paired t-test. The educational presentation will be recorded and emailed to participants within 1 week of intervention to re-watch/review.

DETAILED DESCRIPTION:
The pediatric population faces a public health crisis involving children and adolescents with overweight or obesity. Childhood obesity has become the most disconcerting and predominant pediatric nutritional disorder worldwide. From 2017 to 2018, 19.3% of the children and adolescents in the United States (US) were diagnosed with obesity. Childhood obesity has been linked to psychological conditions such as depression and anxiety. Children that are overweight or obese are more commonly diagnosed with depression than children with a healthy weight. In 2019, 13.6% of children five to seventeen years old received mental health treatment in twelve months, and 8.4% of that population had taken psychotropic medication for their mental health condition.

Healthy lifestyle behaviors impact short and long-term health and quality of life among children with depression. Physical activity (PA), healthy nutritional habits, and maintaining a healthy weight can improve children's quality of life with depression and overweight or obesity. Parents have the most significant influence on their children's health. Thus, family-based intervention studies have been conducted to promote children's healthy lifestyle behaviors. Behavioral interventions that combine nutritional, physical, and behavioral components and parental involvement have proven to be the best and most effective practice for treating and preventing childhood obesity among adolescents 12-17 years old.

Although there is evidence to support that adolescents benefit from peer and family support and group education, there are few in-depth studies documenting lifestyle modifications that can improve this population's overall physical and mental health. Given this lack of implementation into practice, this project aims to improve healthy lifestyle knowledge and behaviors among adolescents with a mental health condition(s) through preventative and detailed nutritional, physical activity, screen time, and sleep education.

This study's purpose is to identify factors that may aid in answering the clinical question: Among adolescents 12-17 years old who are diagnosed with a mental health condition(s), does a family-based educational intervention improve healthy lifestyle knowledge and behaviors, including nutrition, PA, screen time, and sleep? The specific aims are to: Aim 1: To educate adolescents with mental health conditions and their family members about ways to improve healthy lifestyle behaviors. Aim 2: To evaluate an increase in knowledge on healthy lifestyle behaviors after a 45-minute online education session. Aim 3: To evaluate an increase in healthy lifestyle behaviors after the intervention.

ELIGIBILITY:
* Adolescents, 12-17 years old, with a clinical diagnosis of a mental health condition(s) and their parent/legal guardian.
* Examples of eligible diagnosed mental health conditions include major depressive disorder (MDD), generalized anxiety disorder (GAD), attention-deficit disorder (ADD)/ attention deficit hyperactivity disorder (ADHD), bipolar disorder (BPD).
* Adolescents that score below 13 on the World Health Organization (Five) Well-Being Index survey or if the adolescent has answered 0 to 1 to any of the five items, they will not be allowed to complete the REDCap survey or participate in the project unless they are currently enrolled in outpatient mental health services (Ex: counseling, therapy, partial hospitalization).
* Parent(s)/legal guardian(s), 18 years old or older, live with adolescents diagnosed with a mental health condition(s)

Inclusion Criteria:

* Individuals who are not yet adults (Adolescents 12-17 years old)
* With diagnosed mental health condition (ex: Depression, Anxiety, ADD/ADHD) more than one year ago.
* Adolescent eligibility determined with WHO-5 screening prior to pre-intervention survey. o Parent(s)/legal guardian(s), 18 years old or order, live with adolescents diagnosed with mental health condition(s)
* Be able to read/write in English

Exclusion Criteria:

* Children <12 years old or >18 years old
* Children 12-17 that are wards of the state or any other agency, institution, or entity
* Adolescent scoring <13 and not currently enrolled in mental health services, or if the adolescent has answered 0 to 1 to any of the five items, on the WHO-5, and not currently enrolled in mental health services.
* Female participants that report they are pregnant before or after the start of the study will be excluded from the study.
* Parent(s)/legal guardian(s) < 18 years old
* Non-legal guardians

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Livings, Study Chair — Florida State University; Rachel L Sharp, BSN, Principal Investigator — Florida State University
Locations (1):
- Wolfson Children's Hospital- Intensive Outpatient Behavioral Health Program (IOP) and the Partial Hospitalization Program (PHP) and Bridge Program, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Khudairy L, Loveman E, Colquitt JL, Mead E, Johnson RE, Fraser H, Olajide J, Murphy M, Velho RM, O'Malley C, Azevedo LB, Ells LJ, Metzendorf MI, Rees K. Diet, physical activity and behavioural interventions for the treatment of overweight or obese adolescents aged 12 to 17 years. Cochrane Database Syst Rev. 2017 Jun 22;6(6):CD012691. doi: 10.1002/14651858.CD012691. PMID 28639320
- [Background] Barnett ER, Trepman AZ, Fuson HA, Acquilano SC, McLaren JL, Woloshin S, Leyenaar JK. Deprescribing psychotropic medications in children: results of a national qualitative study. BMJ Qual Saf. 2020 Aug;29(8):655-663. doi: 10.1136/bmjqs-2019-010033. Epub 2019 Dec 13. PMID 31836627
- [Background] Bean MK, Caccavale LJ, Adams EL, Burnette CB, LaRose JG, Raynor HA, Wickham EP 3rd, Mazzeo SE. Parent Involvement in Adolescent Obesity Treatment: A Systematic Review. Pediatrics. 2020 Sep;146(3):e20193315. doi: 10.1542/peds.2019-3315. PMID 32839242
- [Background] Blasco BV, Garcia-Jimenez J, Bodoano I, Gutierrez-Rojas L. Obesity and Depression: Its Prevalence and Influence as a Prognostic Factor: A Systematic Review. Psychiatry Investig. 2020 Aug;17(8):715-724. doi: 10.30773/pi.2020.0099. Epub 2020 Aug 12. PMID 32777922
- [Background] Faught EL, Ekwaru JP, Gleddie D, Storey KE, Asbridge M, Veugelers PJ. The combined impact of diet, physical activity, sleep and screen time on academic achievement: a prospective study of elementary school students in Nova Scotia, Canada. Int J Behav Nutr Phys Act. 2017 Mar 9;14(1):29. doi: 10.1186/s12966-017-0476-0. PMID 28274260
- [Background] Gidugu V, Jacobs ML. Empowering individuals with mental illness to develop healthy eating habits through mindful eating: results of a program evaluation. Psychol Health Med. 2019 Feb;24(2):177-186. doi: 10.1080/13548506.2018.1516295. Epub 2018 Aug 31. PMID 30165751
- [Background] Ivey-Stephenson AZ, Demissie Z, Crosby AE, Stone DM, Gaylor E, Wilkins N, Lowry R, Brown M. Suicidal Ideation and Behaviors Among High School Students - Youth Risk Behavior Survey, United States, 2019. MMWR Suppl. 2020 Aug 21;69(1):47-55. doi: 10.15585/mmwr.su6901a6. PMID 32817610
- [Background] Jacka FN. Nutritional Psychiatry: Where to Next? EBioMedicine. 2017 Mar;17:24-29. doi: 10.1016/j.ebiom.2017.02.020. Epub 2017 Feb 21. PMID 28242200
- [Background] Kansra AR, Lakkunarajah S, Jay MS. Childhood and Adolescent Obesity: A Review. Front Pediatr. 2021 Jan 12;8:581461. doi: 10.3389/fped.2020.581461. eCollection 2020. PMID 33511092
- [Background] Leeb RT, Bitsko RH, Radhakrishnan L, Martinez P, Njai R, Holland KM. Mental Health-Related Emergency Department Visits Among Children Aged <18 Years During the COVID-19 Pandemic - United States, January 1-October 17, 2020. MMWR Morb Mortal Wkly Rep. 2020 Nov 13;69(45):1675-1680. doi: 10.15585/mmwr.mm6945a3. PMID 33180751
- [Background] Lindberg L, Hagman E, Danielsson P, Marcus C, Persson M. Anxiety and depression in children and adolescents with obesity: a nationwide study in Sweden. BMC Med. 2020 Feb 21;18(1):30. doi: 10.1186/s12916-020-1498-z. PMID 32079538
- [Background] Loewen OK, Maximova K, Ekwaru JP, Faught EL, Asbridge M, Ohinmaa A, Veugelers PJ. Lifestyle Behavior and Mental Health in Early Adolescence. Pediatrics. 2019 May;143(5):e20183307. doi: 10.1542/peds.2018-3307. Epub 2019 Apr 19. PMID 31004047
- [Background] Merlo CL, Jones SE, Michael SL, Chen TJ, Sliwa SA, Lee SH, Brener ND, Lee SM, Park S. Dietary and Physical Activity Behaviors Among High School Students - Youth Risk Behavior Survey, United States, 2019. MMWR Suppl. 2020 Aug 21;69(1):64-76. doi: 10.15585/mmwr.su6901a8. PMID 32817612
- [Background] Morrison KM, Shin S, Tarnopolsky M, Taylor VH. Association of depression & health related quality of life with body composition in children and youth with obesity. J Affect Disord. 2015 Feb 1;172:18-23. doi: 10.1016/j.jad.2014.09.014. Epub 2014 Sep 23. PMID 25451390
- [Background] Naar S, Ellis D, Idalski Carcone A, Jacques-Tiura AJ, Cunningham P, Templin T, Hartlieb KB, Jen KC. Outcomes From a Sequential Multiple Assignment Randomized Trial of Weight Loss Strategies for African American Adolescents With Obesity. Ann Behav Med. 2019 Aug 29;53(10):928-938. doi: 10.1093/abm/kaz003. PMID 30951586
- [Background] Nigg CR, Wunsch K, Nigg C, Niessner C, Jekauc D, Schmidt SCE, Woll A. Are Physical Activity, Screen Time, and Mental Health Related During Childhood, Preadolescence, and Adolescence? 11-Year Results From the German Motorik-Modul Longitudinal Study. Am J Epidemiol. 2021 Feb 1;190(2):220-229. doi: 10.1093/aje/kwaa192. PMID 33524119
- [Background] Riehm KE, Feder KA, Tormohlen KN, Crum RM, Young AS, Green KM, Pacek LR, La Flair LN, Mojtabai R. Associations Between Time Spent Using Social Media and Internalizing and Externalizing Problems Among US Youth. JAMA Psychiatry. 2019 Dec 1;76(12):1266-1273. doi: 10.1001/jamapsychiatry.2019.2325. PMID 31509167
- [Background] Rippe JM. Lifestyle Medicine: The Health Promoting Power of Daily Habits and Practices. Am J Lifestyle Med. 2018 Jul 20;12(6):499-512. doi: 10.1177/1559827618785554. eCollection 2018 Nov-Dec. PMID 30783405
- [Background] Rodriguez-Ayllon M, Cadenas-Sanchez C, Estevez-Lopez F, Munoz NE, Mora-Gonzalez J, Migueles JH, Molina-Garcia P, Henriksson H, Mena-Molina A, Martinez-Vizcaino V, Catena A, Lof M, Erickson KI, Lubans DR, Ortega FB, Esteban-Cornejo I. Role of Physical Activity and Sedentary Behavior in the Mental Health of Preschoolers, Children and Adolescents: A Systematic Review and Meta-Analysis. Sports Med. 2019 Sep;49(9):1383-1410. doi: 10.1007/s40279-019-01099-5. PMID 30993594
- [Background] Schwartz BS, Glass TA, Pollak J, Hirsch AG, Bailey-Davis L, Moran TH, Bandeen-Roche K. Depression, its comorbidities and treatment, and childhood body mass index trajectories. Obesity (Silver Spring). 2016 Dec;24(12):2585-2592. doi: 10.1002/oby.21627. Epub 2016 Nov 2. PMID 27804225
- [Background] Skelton JA, Buehler C, Irby MB, Grzywacz JG. Where are family theories in family-based obesity treatment?: conceptualizing the study of families in pediatric weight management. Int J Obes (Lond). 2012 Jul;36(7):891-900. doi: 10.1038/ijo.2012.56. Epub 2012 Apr 24. PMID 22531090
- [Background] Williams YV, Cowan PA, Graff JC. Depressive Symptoms, Body Mass Index, and Physical Activity Self-Efficacy in African American Children. J Child Fam Stud. 2020;29(9):2580-2589. doi: 10.1007/s10826-020-01761-x. Epub 2020 Jun 27. PMID 32837149
- [Background] Wu X, Bastian K, Ohinmaa A, Veugelers P. Influence of physical activity, sedentary behavior, and diet quality in childhood on the incidence of internalizing and externalizing disorders during adolescence: a population-based cohort study. Ann Epidemiol. 2018 Feb;28(2):86-94. doi: 10.1016/j.annepidem.2017.12.002. Epub 2017 Dec 11. PMID 29439784
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- See also: Related Info — https://www.healthychildren.org/English/ages-stages/teen/nutrition/Pages/A-Teenagers-Nutritional-Needs.aspx
- See also: Related Info — http://www.healthychildren.org/English/healthy-living/nutrition/Pages/Choose-Water-for-Healthy-Hydration.aspx
- See also: Related Info — https://citl.indiana.edu/teaching-resources/guides/Zoom%20Etiquette.html
- See also: Related Info — https://www.niddk.nih.gov/health-information/weight-management/take-charge-health-guide-teenagers
- See also: Related Info — http://www.myplate.gov
- See also: Related Info — http://health.gov/our-work/nutrition-physical-activity/physical-activity-guidelines/previous-guidelines/2008-physical-activity-guidelines
- See also: Related Info — http://www.census.gov/programs-surveys/nsch/technical-documentation/questionnaires.html
- See also: Related Info — http://www.cdc.gov/healthyyouth/data/yrbs/questionnaires.htm
- See also: Related Info — http://www.corc.uk.net/outcome-experience-measures/the-world-health-organisation-five-well-being-index-who-5/
- See also: Related Info — http://www.psykiatri-regionh.dk/who-5/who-5-questionnaires/Pages/default.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This project enrolled 86 parent-adolescent dyads total (1 parent and 1 adolescent per dyad), and nine parent-adolescent dyads total completed the study. The setting was the Intensive Outpatient Behavioral Health Program (IOP), the Partial Hospitalization Program (PHP), and the Bridge Program at Wolfson Children Hospital in Jacksonville, Fl. Recruitment included posting approved project flyers on social media platforms such as Facebook and Instagram.
Groups:
- Parent-Adolescent Dyad: Each parent-adolescent dyad will receive the intervention (educational program delivered via a 45-minute presentation via Zoom).
  The educational program will promote healthy lifestyle knowledge and behaviors through education evidenced by the CDC, WHO, and the American Academy of Pediatrics. Educational sessions will include the importance of healthy lifestyle modifications in the adolescent population with a mental health condition(s), lifestyle recommendations versus reality, nutrition, physical activity, screen time, and sleep recommendations and guidelines. The educational presentation will include 5-10 minutes of education regarding recommendations versus reality for nutrition, PA, screen time, and sleep, 20-25 minutes of education regarding ways to improve healthy lifestyle knowledge and behaviors, 10 minutes for questions and discussion.
  Zoom Intervention
  * The educational presentation will be recorded and emailed to participants within 1 week of intervention to re-watch/review.
  * Educational sessions will include the importance of healthy lifestyle modifications in the adolescent population with a mental health condition(s), lifestyle recommendations versus reality, nutrition, physical activity, screen time, and sleep recommendations and guidelines.
  * We will compare the effects of an educational program on healthy lifestyle knowledge and behaviors pre-and post-program (after one month) via a REDCap survey for the adolescent and their parent/legal guardian.
Period: Overall Study
Arm/Group | Parent-Adolescent Dyad
Started | 86 (86 total dyads (parent- adolescent dyads). 1 parent and 1 adolescent per dyad.)
Completed | 9 (9 total dyads (parent-adolescent dyads). 1 parent and 1 adolescent per dyad.)
Not Completed | 77

BASELINE CHARACTERISTICS:
Population: Participants (dyads) who completed the pre-survey
Groups:
- Pre-Intervention: Participants (Dyads) who completed the pre-survey
Arm/Group | Pre-Intervention
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants] — Population: The Parent-Adolescent Dyad is presented separately to distinguish parent participants from adolescent participants.
  Participants
    Parents/Legal Guardians: number analyzed (Participants) | 9
    Parents/Legal Guardians: <=18 years | 9
    Parents/Legal Guardians: Between 18 and 65 years | 0
    Parents/Legal Guardians: >=65 years | 0
    Adolescents: number analyzed (Participants) | 9
    Adolescents: <=18 years | 0
    Adolescents: Between 18 and 65 years | 9
    Adolescents: >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 24 [12 to 42]
Age, Customized [Median (Full Range); unit: years] — Population: The Parent-Adolescent Dyad is presented separately to distinguish parent participants from adolescent participants.
  years
    Parent/Legal Guardians: number analyzed (Participants) | 9
    Parent/Legal Guardians | 30 [24 to 42]
    Adolescents: number analyzed (Participants) | 9
    Adolescents | 14 [12 to 17]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Separate parent/legal guardians from adolescents.
  Participants
    Parent/Legal Guardians: number analyzed (Participants) | 9
    Parent/Legal Guardians: Male | 6
    Parent/Legal Guardians: Female | 3
    Adolescents: number analyzed (Participants) | 9
    Adolescents: Male | 6
    Adolescents: Female | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Parent-Adolescent Dyad is presented separately to distinguish parent participants from adolescent participants.
  Participants
    Parents/Legal Guardians: number analyzed (Participants) | 9
    Parents/Legal Guardians: Hispanic or Latino | 3
    Parents/Legal Guardians: Not Hispanic or Latino | 4
    Parents/Legal Guardians: Unknown or Not Reported | 2
    Adolescents: number analyzed (Participants) | 9
    Adolescents: Hispanic or Latino | 6
    Adolescents: Not Hispanic or Latino | 3
    Adolescents: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Parent-Adolescent Dyad is presented separately to distinguish parent participants from adolescent participants.
  Participants
    Parents/Legal Guardians: number analyzed (Participants) | 9
    Parents/Legal Guardians: American Indian or Alaska Native | 0
    Parents/Legal Guardians: Asian | 0
    Parents/Legal Guardians: Native Hawaiian or Other Pacific Islander | 0
    Parents/Legal Guardians: Black or African American | 6
    Parents/Legal Guardians: White | 2
    Parents/Legal Guardians: More than one race | 0
    Parents/Legal Guardians: Unknown or Not Reported | 1
    Adolescents: number analyzed (Participants) | 9
    Adolescents: American Indian or Alaska Native | 0
    Adolescents: Asian | 0
    Adolescents: Native Hawaiian or Other Pacific Islander | 0
    Adolescents: Black or African American | 6
    Adolescents: White | 2
    Adolescents: More than one race | 0
    Adolescents: Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants] — Population: The Parent-Adolescent Dyad is presented separately to distinguish parent participants from adolescent participants.
  Participants
    United States: Parents/Legal Guardians | 9
    United States: Adolescents | 9
Age of Diagnosis for Adolescent Participants Only [Median (Full Range); unit: years] — Parent-reported age that adolescent was diagnosed with mental health condition. Population: The Parent-Adolescent Dyad is presented separately to distinguish parent participants from adolescent participants.
  years
    number analyzed (Participants) | 9
    (all) | 12 [12 to 14]
Parent/Legal Guardian Mood [Median (Full Range); unit: Units on a scale] — Parent-reported current mental health status. Represented on the following 1-5 scale: poor (1), fair (2), good (3), very good (4), excellent (5). Higher values represent better outcomes. The question was copied from the 2021 United States Census Bureau Questionnaire. Population: The Parent-Adolescent Dyad is presented separately to distinguish parent participants from adolescent participants.
  Units on a scale
    number analyzed (Participants) | 9
    (all) | 4 [1 to 5]
Adolescent Weight [Mean (Full Range); unit: lbs] — Population: The Parent-Adolescent Dyad is presented separately to distinguish parent participants from adolescent participants.
  lbs
    number analyzed (Participants) | 9
    (all) | 106 [60 to 150]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Correct Responses for Healthy Lifestyle Behavior Knowledge Survey Questions.
Description: Evaluate knowledge on healthy lifestyle behaviors before and one month after a 45-minute online educational session using a questionnaire (the same questionnaire for before and after intervention).
Time Frame: One Month
Population: This project included nine parent-adolescent dyads. Examples of eligible diagnosed mental health conditions include major depressive disorder (MDD), generalized anxiety disorder (GAD), attention-deficit disorder (ADD)/ attention deficit hyperactivity disorder (ADHD), and bipolar disorder (BPD). Participants' exclusion criteria include children under 12 years old or older than 18 years old. Non-legal guardians were unable to participate in the project.
Measure: Number; unit: percentage of participants
Groups:
- Parent/Legal Guardian (LG) Pre-Intervention Knowledge Changes; Parent/Legal Guardian (LG) Post-Intervention Knowledge Changes: Parent/legal guardians of adolescents 12-17 years old with a clinical diagnosis of a mental health condition(s)
- Adolescent Pre-Intervention Knowledge Changes; Adolescent Post-Intervention Knowledge Changes: Adolescents 12-17 years old with a clinical diagnosis of a mental health condition(s)
Arm/Group | Parent/Legal Guardian (LG) Pre-Intervention Knowledge Changes | Parent/Legal Guardian (LG) Post-Intervention Knowledge Changes | Adolescent Pre-Intervention Knowledge Changes | Adolescent Post-Intervention Knowledge Changes
Number analyzed (Participants) | 9 | 9 | 9 | 9
percentage of participants
  Carbohydrates per day | 33 | 44 | 56 | 33
  Cups of fruit per day | 44 | 67 | 56 | 33
  Cups of Veggies per day | 44 | 56 | 33 | 44
  Cups of water per day | 22 | 44 | 22 | 33
  Healthy snack | 44 | 44 | 44 | 56
  Aerobic Exercise per week | 44 | 44 | 44 | 89
  Example of Aerobic Activity | 33 | 44 | 22 | 56
  Example of BS Activity | 33 | 0 | 0 | 11
  Example of MS Activity | 67 | 33 | 33 | 33
  Exercise per day | 33 | 44 | 22 | 44
  Average screen time | 11 | 22 | 0 | 11
  Recommended screen time | 22 | 11 | 11 | 0
  Reduce screen time | 33 | 11 | 44 | 22
  Recommended hours of sleep | 44 | 11 | 11 | 22
  Risk of poor sleep | 33 | 22 | 33 | 22
  Sleep quality | 67 | 56 | 33 | 56
Statistical Analysis 1: Comparison: Parent/Legal Guardian (LG) Pre-Intervention Knowledge Changes vs Parent/Legal Guardian (LG) Post-Intervention Knowledge Changes; Test type: Other — The descriptive analysis yields frequencies and percentages for categorical variables. The statistical analysis was conducted using IBM SPSS V27.0. We analyzed the percentage of correct responses for knowledge survey questions from pre- and post-intervention survey responses; Participant data was collected from the REDCap pre- and post-intervention questionnaires completed by the adolescents and parents/legal guardians that participated in the project. Data was collected from October to December 2022. The sample size was nine parent-adolescent dyads. Descriptive analysis was used to assess differences in sociodemographic variables, including age, gender, race, material status, employment status, salary, height, and weight. The descriptive analysis yields frequencies and percentages for categorical variables. The statistical analysis was conducted using IBM SPSS V27.0

2. Primary Outcome: Median Score on a Scale of Participants Responses for Healthy Lifestyle Behavior Knowledge Survey Questions
Description: Evaluate healthy lifestyle behaviors before and one month after a 45-minute online educational session using a questionnaire (the same questionnaire for before and after intervention). The scale was adapted from 2021 United States Census Bureau Questionnaire, 2001 PHQ-9, 2021 National Youth Physical Activity and Nutrition Study, and 2021 Youth Risk Behavior Surveillance System Questionnaire. High scores represent better outcomes. The subscale range for each question is as follows: Drink Water 1-7, Eat Breakfast 1-8, Eat dairy products 1-7, eat family dinner 1-8, eat fruit 1-7, eat whole grains 1-7, where do you eat dinner 1-7, eat vegetables 1-7, active 60min/day 1-8, aerobic activity 1-8, Muscle Strengthening Activity 1-8, sports teams 1-4, Bed at Same Time 1-6, Bedtime 7-12, Hours of Sleep 3-12, Nap during day 1-6, restless sleep 1-6, Tired during day 1-6, where do you sleep 1-7, awaken during night 1-6, WHO final score 0-25, afford food 1-3, family dinner 1-8, family exercise 1-8.
Time Frame: One Month
Population: WHO-5 Analysis for Adolescent participants only.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Parent/Legal Guardian (LG) Pre-Intervention Behavioral Changes; Parent/Legal Guardian (LG) Post-Intervention Behavioral Changes: Parent/legal guardians of adolescents 12-17 years old with a clinical diagnosis of a mental health condition(s).
- Adolescent Pre-Intervention Behavioral Changes; Adolescent Post-Intervention Behavioral Changes: Nine adolescents 12-17 years old with a clinical diagnosis of a mental health condition(s)
Arm/Group | Parent/Legal Guardian (LG) Pre-Intervention Behavioral Changes | Parent/Legal Guardian (LG) Post-Intervention Behavioral Changes | Adolescent Pre-Intervention Behavioral Changes | Adolescent Post-Intervention Behavioral Changes
Number analyzed (Participants) | 9 | 9 | 9 | 9
score on a scale
  Drink Water | 5 [1 to 7] | 5 [1 to 7] | 4 [1 to 7] | 5 [1 to 7]
  Eat Breakfast | 5 [1 to 8] | 6 [1 to 8] | 4 [1 to 8] | 5 [1 to 8]
  Eat Dairy Products | 4 [1 to 7] | 6 [1 to 7] | 5 [1 to 7] | 5 [1 to 7]
  Eat Family Dinner | 5 [1 to 8] | 5 [1 to 8] | 5.5 [1 to 8] | 6 [1 to 8]
  Eat Fruit | 4 [1 to 7] | 4 [1 to 7] | 3.5 [1 to 7] | 5 [1 to 7]
  Eat Whole Grains | 5 [1 to 7] | 6 [1 to 7] | 4 [1 to 7] | 5 [1 to 7]
  Where do You Eat Dinner | 4 [1 to 7] | 3.5 [1 to 7] | 2.5 [1 to 7] | 2 [1 to 7]
  Eat Vegetables | 3 [1 to 7] | 4 [1 to 7] | 4 [1 to 7] | 5 [1 to 7]
  Active 60min/day | 4 [1 to 8] | 5 [1 to 8] | 4 [1 to 8] | 5 [1 to 8]
  Aerobic Activity | 5 [1 to 8] | 5 [1 to 8] | 4 [1 to 8] | 5 [1 to 8]
  Muscle Strengthening Activity | 5 [1 to 8] | 6 [1 to 8] | 5 [1 to 8] | 5 [1 to 8]
  Sports Teams | 2 [1 to 4] | 3 [1 to 4] | 2 [1 to 4] | 3 [1 to 4]
  Bed at Same Time | 3 [1 to 6] | 3 [1 to 6] | 4 [1 to 6] | 4 [1 to 6]
  Bedtime | 8 [7 to 12] | 8 [7 to 12] | 8 [7 to 12] | 8 [7 to 12]
  Hours of Sleep | 6 [3 to 12] | 6 [3 to 12] | 6 [3 to 12] | 7.5 [3 to 12]
  Nap During Day | 3 [1 to 6] | 3 [1 to 6] | 3.5 [1 to 6] | 4 [1 to 6]
  Restless Sleep | 3 [1 to 6] | 4 [1 to 6] | 4 [1 to 6] | 4 [1 to 6]
  Tired During Day | 4 [1 to 6] | 4 [1 to 6] | 4 [1 to 6] | 4 [1 to 6]
  Where do You Sleep | 2 [1 to 7] | 2 [1 to 7] | 2 [1 to 7] | 1 [1 to 7]
  Awaken During Night | 4 [1 to 6] | 4 [1 to 6] | 3.5 [1 to 6] | 4 [1 to 6]
  WHO-5 Final Score: number analyzed (Participants) | 0 | 0 | 9 | 9
  WHO-5 Final Score |  |  | 13 [0 to 25] | 16 [0 to 25]
  Afford Food | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
  Family Dinner | 4 [1 to 8] | 5 [1 to 8] | 4.5 [1 to 8] | 6 [1 to 8]
  Family Exercise | 5 [1 to 8] | 5 [1 to 8] | 3 [1 to 8] | 5 [1 to 8]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Parent/Legal Guardian (LG) Pre-Intervention Knowledge Changes | Parent/Legal Guardian (LG) Post-Intervention Knowledge Changes | Adolescent Pre-Intervention Knowledge Changes | Adolescent Post-Intervention Knowledge Changes
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2022-11-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT05675020/Prot_SAP_004.pdf
  • Informed Consent Form: Adult- General Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT05675020/ICF_001.pdf
  • Informed Consent Form: Adolescent 14-17yr - Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT05675020/ICF_002.pdf
  • Informed Consent Form: Child 7-13yr- Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT05675020/ICF_003.pdf